CLINICAL TRIAL: NCT04291209
Title: Intratympanic N-Acetylcysteine (NAC) Injections for Prevention of Cisplatin-induced Ototoxicity in Head and Neck Cancer Patients: A Multi-centre Phase II Randomized Controlled Trial.
Brief Title: Intratympanic N-Acetylcysteine for Prevention of Cisplatin-induced Ototoxicity.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Toronto Sunnybrook Regional Cancer Centre (Other); London Regional Cancer Program, Canada (Other)
Responsible Party: Principal Investigator, Dr. Trung Le, Trung N. Le MD PhD, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1819
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Ototoxic Hearing Loss
Keywords: Hearing Loss; Deafness; Cisplatin-induced Ototoxicity; Sensorineural hearing loss; Ear diseases; Antioxidant; N-acetyl cystein
MeSH Terms: conditions — Hearing Loss; Deafness; Hearing Loss, Sensorineural; Ear Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm with Intratympanic NAC injection (Active Comparator): One ear will be randomly chosen for the experimental treatment and receive intratympanic NAC injections 60 minutes prior to their scheduled chemotherapy sessions
  Interventions: Drug: N-Acetyl Cysteine
- Control arm with No injection (No Intervention): The control ear will not receive any injections

INTERVENTIONS:
Drug: N-Acetyl Cysteine — One ear will be randomly chosen for the experimental treatment of intratympanic NAC. The other ear will serve as the control ear which will not receive any injection.
  Other Names: NAC
  Arms: Experimental arm with Intratympanic NAC injection

SUMMARY:
Although many intratympanic agents have been attempted, N-Acetylcysteine (NAC) appears to be the most promising and is a powerful, commonly used anti-oxidant. The goal of this prospective phase 2 randomized controlled trial is to determine the optimal dosage and effectiveness of intratympanic NAC injection in reducing hearing loss in head & neck cancer patients receiving cisplatin chemotherapy with curative intent.

DETAILED DESCRIPTION:
A prospective randomized controlled trial phase 1 using a standard 3+3 design, followed by a randomized controlled phase 2 to determine dosage, safety, and efficacy of intratympanic NAC to treat hearing loss in head & neck patients receiving high-dose cisplatin chemotherapy. Participants will complete various pre-treatment hearing tests. One ear will be randomly chosen for the experimental treatment and the other ear will serve as the control ear. Participants will receive intratympanic NAC injections 60 minutes prior to their scheduled chemotherapy sessions in the experimental ear. The control ear will not receive any injection. Follow up hearing tests will be performed 2 months following completion of their primary cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage head and neck cancer
* Receiving high dose systemic cisplatin (100mg/m2) with concurrent radiation therapy as part of their curative intent treatment
* Willing to provide informed consent
* ECOG performance status 0-2
* Histological confirmation of squamous cell carcinoma

Exclusion Criteria:

* Age less than 18
* Metastatic disease
* Tympanic membrane perforation or the presence of tympanostomy tubes as this may impact the retention and absorption of NAC when inserted into the middle ear
* Preexisting severe to profound sensorineural hearing loss (unilateral or bilateral)
* Pretreatment interaural discrepancy of greater than 10dB at three frequencies
* History of Meniere's or fluctuating hearing loss
* Previous hypersensitivity to NAC
* Patient unable to follow the protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Determination of a safe and tolerable dosage for intratympanic NAC injection | Within 1 day
  The primary end-point of the phase 1 part of this study is the safety and tolerability of intratympanic NAC injections, by determining the causality of adverse events and serious adverse events and grading according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v.5.0
Improvement in hearing threshold with intratympanic NAC injection | Within 2 months
  The primary outcome measure of this study will be a comparison of hearing loss between the control and NAC-injected ears. More specifically, each ear will be scored as having hearing loss if there is a greater than 10dB hearing loss in three contiguous frequencies. This will be measured via threshold hearing tests.

SECONDARY OUTCOMES:
Improvement in hearing quality with intratympanic NAC injection | Within 2 months
  The secondary outcome measure of this study will be a comparison of hearing discrimination, subjective tinnitus, otoacoustic emission, speech spatial and quality of hearing between the control and NAC-injected ears.

CONTACTS AND LOCATIONS:
Overall Officials: Trung N Le, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No